CLINICAL TRIAL: NCT06749691
Title: Study of Liposomal Irinotecan Combined with Apatinib in the Treatment of Extensive Stage Small Cell Lung Cancer After First-line Progression
Brief Title: Liposomal Irinotecan and Apatinib in ES-SCLC
Acronym: LIAES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhong Xian, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAH-2024-0770
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: Small Cell Lung Cancer; Liposomal Irinotecan; Apatinib
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal Irinotecan and Apatinib (Experimental)
  Interventions: Drug: Liposomal Irinotecan and Apatinib

INTERVENTIONS:
Drug: Liposomal Irinotecan and Apatinib — Liposomal Irinotecan in Combination With Apatinib

SUMMARY:
The purpose of this study is to observe the efficacy and safety of liposomal irinotecan combined with apatinib in the treatment of extensive stage small cell lung cancer progressed from first-line regimen.

DETAILED DESCRIPTION:
Small cell lung cancer is a highly invasive neuroendocrine tumor characterized by high malignancy and rapid proliferation. Although most patients with extensive SCLC are sensitive to first-line treatments such as etoposide combined with platinum and immunotherapy, most patients experience disease progression again after first-line treatment. Therefore, extending the survival time of patients and improving their quality of life have become key issues in the second-line treatment of SCLC. The current guidelines for second-line treatment of SCLC recommend monotherapy, including topotecan, irinotecan, etc. However, the available options have poor efficacy and are prone to drug resistance. Irinotecan liposomes improve drug stability and prolong circulation time through liposome encapsulation, and target tumor tissues through high permeability and long retention effects, with the expected effect of reducing toxicity and increasing efficacy. Apatinib is a small molecule tyrosine kinase inhibitor that selectively inhibits vascular endothelial growth factor receptors to achieve anti angiogenic and anti-tumor effects. It has been proven to have positive therapeutic effects in multiple types of cancer, including SCLC. At present, the combination mode of chemotherapy and anti-angiogenic drugs has been explored in various tumors, and the results show that this mode has drug synergistic effects, which can significantly improve the efficacy of anti-tumor treatment. Therefore, exploring the efficacy, safety, and mechanism of liposomal irinotecan combined with apatinib is of great clinical and theoretical significance for the refractory tumor population of extensive stage small cell lung cancer with first-line treatment progress.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-75 years;
2. Expected survival period ≥ 12 weeks;
3. At least one measurable lesion (according to RECIST V 1.1);
4. For patients who have failed first-line or second-line treatment.

Exclusion Criteria:

1. Have received any systemic treatment targeting VEGF or VEGFR in the past, such as treatment with anti angiogenic drugs such as ranibizumab, fipronib, apatinib, anlotinib, lenvatinib, sunitinib, sorafenib.
2. Active or uncontrolled severe infection (CTCAE 5.0 ≥ 2) and/or antibiotic treatment within 2 weeks prior to enrollment;
3. There are multiple factors that affect the absorption of oral medication, such as inability to swallow, nausea and vomiting, chronic diarrhea, and intestinal obstruction;
4. Those deemed unsuitable for inclusion by doctors;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival rate at 6 months | From enrollment at 6 months
  Progression-Free-Survival rate at 6 months from enrollment

SECONDARY OUTCOMES:
ORR | From enrollment to the end of treatment at 6-8 weeks
  Overall Response Rate
mPFS | From enrollment to the end of treatment at 6-8 weeks
  median Progression-Free-Survival time
mOS | From enrollment to the end of life at 3 months
  median Overall Survival time

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No